CLINICAL TRIAL: NCT06712277
Title: The Effect of Video Education on Adaptation to the Procedure of Patients and Caregivers Who Underwent Gastrostomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melike YAZAR (Other)
Collaborators: Halic University (Other)
Responsible Party: Sponsor-Investigator, Melike YAZAR, Specialist Nurse, Beykoz State Hospital
Organization: Beykoz State Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Beykoz State Hospital; Higher Education Institution (Other: Higher Education Institution)
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Having a Percutaneous Endoscopic Gastrostomy
Keywords: patients; percutaneous endoscopic gastrostomi; education

STUDY DESIGN:
Intervention Model Description: It was planned as a single-group quasi-experimental study to determine the effect of training on patient and caregiver compliance with gastrostomy and the caregiver's gastrostomy care skills.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients and caregivers who underwent percutaneous endoscopic gastrostomy for the first time (Experimental)
  Interventions: Other: Video training

INTERVENTIONS:
Other: Video training — After the procedure, caregivers will be trained on tube care and patient feeding by demonstrating and performing the procedure on an iPad.

SUMMARY:
This study will be conducted to investigate the effects of video training given to caregivers of patients who underwent percutaneous endoscopic gastrostomy on the compliance of patients and caregivers to gastrostomy. A single-group quasi-experimental study was planned to determine the effect of training on the compliance of patients and caregivers to gastrostomy and the caregiver's gastrostomy care skills. The universe of the study will consist of caregivers who met the inclusion criteria for the study in which gastrostomy procedure was performed for the first time at Beykoz State Hospital between the dates of September 1, 2024 and March 31, 2026. G*Power power analysis was performed to determine the sample size. According to Cohen's effect size coefficients; according to the calculation made assuming that it will have a large effect size (d=0.8), it was decided that there should be at least 20 people with α=0.05 level, 95% power; considering the losses, it was decided to include 25 people in the study. Statistical Package for the Social Sciences 26 program will be used for statistical analyses of the data obtained from the study. While evaluating the study data, descriptive statistical methods (mean, standard deviation, median, frequency and ratio) as well as Shapiro Wilks test and Box Plot graphics will be used in the evaluation of the distribution of the data. Student t test, Oneway Anova test will be used in the evaluation of variables showing normal distribution and Bonferroni test will be used in the determination of the group causing the difference. Paired Samples t test will be used in the evaluations within the groups. Mann Whitney U test, Kruskal Wallis test will be used in the evaluations of variables not showing normal distribution and Dunn test will be used in the determination of the group causing the difference. Wilcoxon Signed Rank test will be used in the evaluations within the groups. Pearson or Spearman's correlation analysis, linear regression modeling will be done in the evaluation of variables. Chi-Square test and Fisher's Exact test will be used in the comparison of qualitative data. The results will be evaluated at a confidence interval of 95% and significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Having undergone percutaneous endoscopic gastrostomy for the first time. Not having cancer. -

Exclusion Criteria:

Being over 18 years old, Being able to communicate in Turkish, Being able to read and write, The caregiver will be involved in the percutaneous endoscopic gastrostomy care of their patient.

Not being a healthcare professional.

-

Max Age: 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
caregiver gastrostomy compliance form | 1-2 month
  It consists of 5 questions that allow the caregiver to express their concerns and troubles while feeding, dressing the tube, giving medication, positioning, and giving body care/bathing to the patient due to the procedure with a value between 0 and 10. The caregiver can get the lowest score from this form: 0, the highest score: 50. A score of 0 from the Caregiver Gastrostomy Adaptation Form indicates that there is no adaptation to gastrostomy, and a score of 50 indicates that there is adaptation to gastrostomy. The form will be finalized after receiving the opinions of 10 experts on the form.

SECONDARY OUTCOMES:
Care Skills Assessment Form | 1-2 month
  It consists of 29 questions measuring care skills, which was created by the researcher in line with the literature in order to evaluate the effectiveness of the training given to the caregivers of the patient with percutaneous endoscopic gastrostomy. The first 27 questions in the care skill evaluation form are worth Yes: 2 points, No: 0 points, Partially: 1 point. 54 points were determined as the highest skill score, 0 points as the lowest skill score. Questions 28 and 29 were created for the evaluation of dressing. The Caregiver Skill Evaluation Form will be filled out by the researcher during the home visit by observing the caregivers on the 14th and 30th day follow-ups. The form will be finalized after receiving the opinions of 10 experts on the form.

OTHER OUTCOMES:
Patient Gastrostomy Compliance Form | 1-2 month
  It was created by the researcher to question the complications that may occur in the patient, the reason for hospitalization and readmission. The form created by the researcher in line with the literature consists of 18 questions (Kahveci, 2020; Torun, 2023). It will be scored as Yes: 1, No: 0. High scores will indicate incompatibility. The form will be finalized after receiving the opinions of 10 experts on the form.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Yazar, Principal Investigator — Beykoz State Hospital Surgical Service Nurse
Locations (1):
- Beykoz State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data collection phase has not been completed yet.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT06712277/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT06712277/ICF_001.pdf